CLINICAL TRIAL: NCT04497233
Title: Prediction Model of Benign and Malignant Peripheral Pulmonary Lesions Based on Image of Radial Endobronchial Ultrasound
Brief Title: Prediction Model of Peripheral Pulmonary Lesions Based on R-EBUS Image
Acronym: R-EBUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director,Endoscope Department,Shanghai Chest Hospital, Shanghai Chest Hospital
Other Study IDs: SHCHE202001
Record Dates: First submitted 2020-07-19; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Diagnoses Disease
Keywords: R-EBUS image; Deep learning; Peripheral pulmonary lesions; Prediction model; Diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospectively validation group: Two diagnosis methods will be used in the prospective validation section, one is traditional qualitative and quantitative method, the other is artificial intelligence prediction model based on videos to compare the diagnostic efficacy.

SUMMARY:
Peripheral pulmonary lesions(PPLs) have a wide spectrum of diseases, and the diagnosis will affect the treatment strategy and prognosis. Radial endobronchial ultrasound (R-EBUS) can be used for non-invasive diagnosis of PPLs, and the supplement pathological diagnosis results of EBUS-TBLB, which has important clinical application value. This project intends to select representative images from R-EBUS dynamic videos for qualitative and quantitative analysis, to establish and verify the diagnostic evaluation system of R-EBUS forPPLs. Then build 1,000 R-EBUS image databases of PPLs, train deep learning networks for automatic extraction and diagnosis of target areas, and automatically extract representative images from videos to establish a benign and malignant prediction model of PPLs. We will provide reliable theoretical basis for the diagnosis of PPLs, and optimize the diagnosis and treatment method.The network would be prospectively verified through 300 R-EBUS images from multi centers.

DETAILED DESCRIPTION:
PPLs are lesions at tertiary bronchus and above. The lesion cannot be seen by conventional bronchoscopy and the diagnosis will affect the treatment strategy and prognosis. R-EBUS can be used for non-invasive diagnosis of PPLs, and the supplement pathological diagnosis results of EBUS-TBLB. During the procedure, target PPLs are examined by ultrasound host (EU-ME2, Olympus, Tokyo, Japan) equipped with Doppler function and ultrasound probe . The bronchoscope reaches the distal as far as possible according to the predetermined position on chest CT or positron emission tomography-computed tomography (PET-CT) . The R-EBUS probe is inserted into the working channel of the bronchoscope, and gradually approaches the target PPL to obtain R-EBUS image. According to the characteristics such as within or adjacent to image, the probe scan the lesion from the near end to the far end and record the video. The recording time is required longer than 10 seconds. After selecting a typical R-EBUS image, freeze the image and take a screenshot. The long and short diameter of the lesion will be measured. This project includes three parts: preliminary construction and evaluation of R-EBUS image system for benign and malignant PPLs, construction of R-EBUS artificial intelligence prediction model and multi-center prospective validation of the prediction model. A total of 1000 patients will be enrolled to construct diagnostic model and 300 are enrolled to verify the diagnostic effiency.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with PPLs in Chest CT or PET / CT;
2. Chest CT or PET / CT shows PPLs with diameter greater than 8 mm;
3. Patients agree to perform EBUS-TBLB and sign the informed consent.

Exclusion Criteria:

1. Thin-layer Chest CT or PET / CT indicates lack of bronchial access to PPLs;
2. Patients refuse to participate in this clinical trial;
3. Patients with severe cardiopulmonary dysfunction or other indications that not allowed for bronchoscopy;
4. Visible lesions in the lumen during conventional bronchoscopy;
5. Patients have other related contraindications of bronchoscopy;
6. Patients have other reasons unfit for this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population of this study are those who meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy of R-EBUS prediction model. | 18 months
  Diagnostic efficacy includes sensitivity, specificity, positive predictive value, negative predictive value and diagnostic accuracy

SECONDARY OUTCOMES:
Diagnostic efficacy of traditional qualitative and quantitative methods | 18 months
  Diagnostic efficacy includes sensitivity, specificity, positive predictive value, negative predictive value and diagnostic accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, PhD, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided